CLINICAL TRIAL: NCT02795949
Title: Randomized, Multicenter, Phase III, Controlled Clinical Trial, to Demonstrate the no Inferiority of Reduced Antibiotic Treatment vs a Broad Spectrum Betalactam Antipseudomonal Treatment in Patients With Bacteremia by Enterobacteriaceae
Brief Title: Study on Reduced Antibiotic Treatment vs Broad Spectrum Betalactam in Patients With Bacteremia by Enterobacteriaceae
Acronym: SIMPLIFY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Spanish Network for Research in Infectious Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIMPLFY
Record Dates: First submitted 2016-04-01; First posted 2016-06-10 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Enterobacteriaceae Infections
Keywords: Enterobacteriaceae; Bacteremia; Escalation; Bacterial resistance; Bloodstream infection; Recurrence
MeSH Terms: conditions — Enterobacteriaceae Infections; Bacteremia; Sepsis; Recurrence | interventions — Ampicillin; Trimethoprim, Sulfamethoxazole Drug Combination; Cefuroxime; Amoxicillin-Potassium Clavulanate Combination; Ciprofloxacin; Ertapenem; Piperacillin, Tazobactam Drug Combination; Meropenem; Imipenem; Aztreonam; Ceftazidime; Cefepime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antipseudomonal beta-lactam antibiotic (Experimental): 1. Ampicillin 2g IV/6h
  2. Trimethoprim/sulfamethoxazole 160/800 mg IV/8 -12h
  3. Cefuroxime 750-1000 mg IV/8h
  4. Cefotaxime 1-2g IV/8h ó ceftriaxone 1 g/12-24h
  5. Amoxicillin/clavulanate 1000/125 mg IV/8h
  6. Ciprofloxacin 400 mg IV/12h
  7. Ertapenem 1-2g/24h.
  Interventions: Drug: Antipseudomonal beta-lactam antibiotic
- De-escalation(short-spectrum antibiotic) (Active Comparator): * Piperacillin/tazobactam 4/0.5 g IV/8h
  * Meropenem 1-2 g IV/8h
  * Imipenem 0.5 g IV/6h - 1g IV/6h
  * Aztreonam 1-2 g IV/8h
  * Ceftazidime 1-2 g IV/8h
  * Cefepime 2 g IV/8-12h
  Interventions: Drug: De-escalation(short-spectrum antibiotic)

INTERVENTIONS:
Drug: Antipseudomonal beta-lactam antibiotic — Pharmaceutical form: solution for infusion
  Other Names: Ampicillin; Trimethoprim/sulfamethoxazole; Cefuroxime; Amoxicillin/clavulanate; Ciprofloxacin; Ertapenem
  Arms: Antipseudomonal beta-lactam antibiotic
Drug: De-escalation(short-spectrum antibiotic) — Pharmaceutical form: solution for infusion
  Other Names: Piperacillin/tazobactam; Meropenem; Imipenem; Aztreonam; Ceftazidime; Cefepime
  Arms: De-escalation(short-spectrum antibiotic)

SUMMARY:
The continuous increase in the bacterial resistance rate and the slow arrival of new therapeutic options have turned into an antibiotic crisis. One of the strategies proposed by stewardship programs to try to change this situation described worldwide is the use of antibiotics with the lowest possible antimicrobial spectrum.

Enterobacteriaceae bacteremia is a good example of how this strategy would be applied. The empirical treatment of nosocomial bacteremia by Enterobacteriaceae comprises in several cases one or two antibiotics with antipseudomonal activity, being much less common than desirable a subsequent change to narrower spectrum antibiotics based on susceptibility data ("de escalation"). This is because the safety of de escalation is based only on expert advice and some observational studies, so their efficacy and safety is questioned by many clinicians and therefore its use is lower than desired. In fact, a recent systematic review of the Cochrane Library concluded that randomized studies to support this practice are needed. Investigators propose a "real clinical practice-based" randomized trial to compare the efficacy and safety of continuing with an antipseudomonal agents vs. de-escalation according to a pre-specified rule, in patients with bacteraemia due to Enterobacteriaceae.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old hospitalized patients with bacteremia from any source with isolation of an enterobacteria in blood cultures.
2. Active empiric treatment with antipseudomonal betalactamic at 48 hours from the symptoms of sepsis and the blood culture.The patient could have received any other type of antibiotic therapy up to 24 hours after blood extraction.
3. Microorganism susceptible at least one treatment from the experimental arm.
4. Patients with intravenous treatment at least 3 days from the randomization o 5 days from the initial blood culture.
5. Patients to sign the informed consent form.

Exclusion Criteria:

1. Palliative care or life expectance < 90 days.
2. Pregnancy or lactation period.
3. To isolate the Extended-spectrum β-lactamases producing Enterobacteriaceae
4. Late randomization >48 hours after the enterobacteriaceae blood culture´s identification
5. Severe neutropenic (< 500 céls/mm3) at the randomization.
6. Treatment of infection > 28 days (endocarditis and osteomyelitis) or meningitis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Clinical cure at day 3-5 after treatment. | Day 3-5 after end of treatment.
  Clinical cure: complete resolution of infection symptoms (bacteremia) present at the day on which the assessment is done and patient is alive.

SECONDARY OUTCOMES:
Early clinical and microbiological response. | After 5 days of treatment
  The infection was completely resolved after 5 days of treatment (patients without infection symptoms and a negative blood culture).
Late clinical and microbiological response. | Day 60
  The infection was completely resolved at day 60 (patients without infection symptoms)
Mortality | At 7,14 and 30 days
  Death for any reason
Length of hospital stay | At 7,14 and 30 days
  Defined as the from admission to hospital discharge
Recurrences (relapse or reinfection) rate | Day 60 after treatment
Safety of antibiotic treatment | 60 days
  Gathering any related adverse event from the informed consent form signature up to 60 days
Impact of the study treatment on intestinal microbiota | Screening, Day 7-14, Day 12-21, Day 30
  Effect of study treatment on colonization of the intestinal tract with multi drug resistant gram negative bacilli
Treatment duration. | It is not allowed treatment duration more than 28 days
  Evaluate the study treatment duration.
Secondary infections. | 60 days
  Evaluate the development of secondary infections other than the initial bacteremia.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Eduardo Lopez Cortes, MD, PhD, Principal Investigator — Universitary Hospital Virgen Macarena
Locations (21):
- Spain (21):
  - Cruces Hospital, Barakaldo, Basque Country
  - Jerez de la Frontera Hospital, Jerez de la Frontera, Cádiz
  - La Línea de La Concepción Hospital, La Línea de la Concepción, Cádiz
  - University Hospital Donostia, Donostia / San Sebastian, Gipúzcoa
  - San Juan de Dios del Aljarafe Hospital, Bormujos, Sevilla
  - La Coruña Hospital, A Coruña
  - University General Hospital of Alicante, Alicante
  - University Hospital Mutua de Tarrasa, Barcelona
  - University Hospital of Bellvitge, Barcelona
  - University Hospital Puerta del Mar, Cadiz
  - Puerto Real Hospital, Cadiz
  - Universitary Hospital of Leon, León
  - University Hospital La Princesa, Madrid
  - University Hospital La Paz, Madrid
  - Universitary Hospital of Orense, Ourense
  - Son Espases Hospital, Palma de Mallorca
  - University Clinic of Navarra, Pamplona
  - University Hospital Marqués de Valdecilla, Santander
  - University Hospital Virgen Macarena, Seville
  - Universitary Hospital of Vigo, Vigo
  - University Hospital of Zaragoza, Zaragoza

REFERENCES:
- [Derived] Lopez-Cortes LE, Delgado-Valverde M, Moreno-Mellado E, Goikoetxea Aguirre J, Guio Carrion L, Blanco Vidal MJ, Lopez Soria LM, Perez-Rodriguez MT, Martinez Lamas L, Arnaiz de Las Revillas F, Arminanzas C, Ruiz de Alegria-Puig C, Jimenez Aguilar P, Del Carmen Martinez-Rubio M, Saez-Bejar C, de Las Cuevas C, Martin-Aspas A, Galan F, Yuste JR, Leiva-Leon J, Bou G, Capon Gonzalez P, Boix-Palop L, Xercavins-Valls M, Goenaga-Sanchez MA, Anza DV, Caston JJ, Rufian MR, Merino E, Rodriguez JC, Loeches B, Cuervo G, Guerra Laso JM, Plata A, Perez Cortes S, Lopez Mato P, Sierra Monzon JL, Rosso-Fernandez C, Bravo-Ferrer JM, Retamar-Gentil P, Rodriguez-Bano J; SIMPLIFY study group. Efficacy and safety of a structured de-escalation from antipseudomonal beta-lactams in bloodstream infections due to Enterobacterales (SIMPLIFY): an open-label, multicentre, randomised trial. Lancet Infect Dis. 2024 Apr;24(4):375-385. doi: 10.1016/S1473-3099(23)00686-2. Epub 2024 Jan 9. PMID 38215770
- [Derived] Lopez-Cortes LE, Rosso-Fernandez C, Nunez-Nunez M, Lavin-Alconero L, Bravo-Ferrer J, Barriga A, Delgado M, Lupion C, Retamar P, Rodriguez-Bano J; SIMPLIFY Study Group. Targeted simplification versus antipseudomonal broad-spectrum beta-lactams in patients with bloodstream infections due to Enterobacteriaceae (SIMPLIFY): a study protocol for a multicentre, open-label, phase III randomised, controlled, non-inferiority clinical trial. BMJ Open. 2017 Jun 9;7(6):e015439. doi: 10.1136/bmjopen-2016-015439. PMID 28601833
- See also: Spanish Network for Research in Infectious Diseases (Red Española de Investigación en Patología Infecciosa) — http://www.reipi.org/